CLINICAL TRIAL: NCT05513079
Title: The Effect of Positive Psychotherapy-Based Counseling (PPT) on Anxiety Levels and Quality of Life of Patients With Chronic Urticaria
Brief Title: Positive Psychotherapy-Based Counseling (PPT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Eda Albayrak, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ErciyesUnı
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Chronic Urticaria; Anxiety
Keywords: Positive Psychotherapy (PPT); Chronic Urticaria; Anxiety; Life quality
MeSH Terms: conditions — Chronic Urticaria; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Individuals in the control group agreed to participate in the study after being explained about the research.
  Verbal and written consent will be obtained from individuals who do so. Initial interview with individuals who agreed to participate in the study Introductory Information Form, Trait Anxiety Scale, Dermatological Quality of Life Scale, Urticaria Activity Score will be applied. Patients in this group have routine chronic No application will be made other than the treatment of urticaria. 5 months after the pre-test Trait State Anxiety Scale, Dermatological Quality of Life Scale, Urticaria Activity Score will be applied. After the study is completed, individuals in the control group can also request it.
  counseling will be provided.
- Intervention Group (Experimental): Positive psychotherapy counseling sessions, specialist psychiatry who completed positive psychotherapy training will be done by the nurse. The first one face-to-face with each individual in the intervention group. A total of 8 sessions will be held, theothers being online. Audio and video with attendees Other sessions will be completed through a program that allows sharing (WhatsAap, zoom etc.). Each session will be applied once a week, lasting 45-50 minutes. Interviews with individuals No audio or video recording will be taken during the recording.
  Interventions: Behavioral: Positive Psychotherapy Based Counseling

INTERVENTIONS:
Behavioral: Positive Psychotherapy Based Counseling — The main purpose in Positive Psychotherapy is to develop the individual's main capacities. and to maintain balance in the four areas of life (body, success, relationships and future) in daily life. to help provide. The essence of Positive Psychotherapy is a five-step process: 1. Observation/distance phase, 2. Inventory phase, 3. Situational encouragement phase, 4. Verbalization phase, 5. Expanding the objectives phase. Shaping five-step model therapy It is a helpful guide.
  Other Names: Positive Psychotherapy (PPT)
  Arms: Intervention Group

SUMMARY:
Chronic urticaria is a condition that impairs the patient's quality of life, interferes with routine daily activities, and is often associated with anxiety.

It constitutes a significant burden associated with psychiatric comorbidities such as Fundamentals of Positive Psychotherapy (PPT) The aim is to help the individual to develop his/her core capacities and in his/her daily life in four areas of life (body, success, relationships and the future) to help them achieve balance. In patients with chronic urticaria, especially problems with the body occur and this can affect other areas of life. Literature When examined, it is seen that psychological interventions in chronic urticaria are very few and in ancient times.

In addition, it is recommended that psychological interventions based on conversation should be performed with these patients. PPT, conversational and balancing the dimensions of "body, achievement, relationships and future" It is a working approach. Body and future in the disease process of chronic urticaria patients Considering that there is a balance change in the dimensions of the PPT, it will contribute to the literature.

is considered. Intervention Group Positive psychotherapy counseling sessions, specialist psychiatry who completed positive psychotherapy training will be done by the nurse. Contact information of the volunteers will be obtained at the outpatient clinic and individuals will be randomized.

will be divided into intervention and control groups. The first one face-to-face with each individual in the intervention group.

A total of 8 sessions will be held, the others being online. Individuals who agreed to participate in the study were first Introductory Information Form, Continuity Anxiety Scale, face-to-face during the interview, Dermatological Quality of Life Scale, Urticaria Activity Score will be applied. Audio and video with volunteers Other sessions will be completed through a program that allows sharing (WhatsAap, zoom etc.).

Each session will be applied once a week, lasting 45-50 minutes. Interviews with individuals No audio or video recording will be taken during the recording. This information was given to the volunteers included in the intervention group.

will be announced before the meeting begins. After the eight-week counseling program 3 months later (pretest-posttest when including the 8-week program to be applied after the pretest) There will be a total of 5 months between Project Title Positive Psychotherapy Based Counseling (PPT) Diagnosed with Chronic Urticaria Anxiety Levels of Patients and Its Effect on Quality of Life Project Coordinator Assoc. Dr. Nuray SIMSEK Researcher(s) Res. See. Eda Albayrak Project Type Ph.D. Thesis Project Project Group ( ) Science and Engineering Sciences ( X) Medicine and Health Sciences ( ) Social Sciences Writing fields can be extended as needed Quality Scale, Urticaria Activity Score will be applied. Control Group Individuals in the control group agreed to participate in the study after being explained about the research.

Verbal and written consent will be obtained from individuals who do so. Initial interview with individuals who agreed to participate in the study Introductory Information Form, Trait Anxiety Scale, Dermatological Quality of Life Scale, Urticaria Activity Score will be applied. Patients in this group are routinely chronically ill.

No application will be made other than the treatment of urticaria. 5 months after the pre-test Trait State Anxiety Scale, Dermatological Quality of Life Scale, Urticaria Activity Score will be applied. After the study is completed, individuals in the control group can also request it.

counseling will be provided.

ELIGIBILITY:
Inclusion Criteria:

Those diagnosed with chronic urticaria Those between the ages of 18-50 Patients without cognitive clouding Anyone with a smartphone/computer who can participate in positive psychotherapy (PPT) sessions Patients who can speak Turkish Patients without hearing and vision problems will be included in the study.

Exclusion Criteria:

Those over 50 or under 18 Having a psychiatric illness and taking medication Have any other chronic disease Those with hearing, vision, speech and cognitive dysfunction, Those who do not speak Turkish Writing fields can be extended as needed Patients who do not accept the procedure will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
State Trait Anxiety Scale | Timeframe: Change: [Timeframe: 5 months: Initial interview (Time 1), 5 months later (Time 2)]
  The total score obtained from both scales varies between 20 and 80. big score high anxiety A low score indicates a low level of anxiety.
Dermatological Quality of Life Scale | Timeframe: Change: [Timeframe: 5 months: Initial interview (Time 1), 5 months later (Time 2)]
  The total score obtained varies between 0-44, and the high total score is associated with the survival of the patients.
  indicates a decrease in quality.

SECONDARY OUTCOMES:
Urticaria Activity Score | Timeframe: Change: [Timeframe: 5 months: Initial interview (Time 1), 5 months later (Time 2)]
  Scoring is evaluated between 0-42 points. Seven-day urticaria activity score; Total (minimum 0-maximum 42) UAS7 score of ≤6 is well-controlled, between 7-15 is mild, 16-27 Between 28 and 42 is considered as moderate urticaria.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes Universty, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided